CLINICAL TRIAL: NCT04461717
Title: Prospective Observational Study of Procedures With MicroNet Covered Stent Use to Treat Increased Risk Lesions in Arterial Locations Beyond the Carotid Bifurcation - FLOW-Guard Study
Brief Title: Micronet Covered Stent in in Arterial Locations Beyond the Carotid Bifurcation - FLOW-Guard Study
Acronym: FLOW-Guard
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: John Paul II Hospital, Krakow (Other)
Responsible Party: Sponsor
Other Study IDs: FLOW-Guard
Record Dates: First submitted 2020-06-08; First posted 2020-07-08 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MicroNet covered stenting (interventional): MicroNet covered stent implantation for increased risk arterial lesions beyond the carotid bifurcation
  Interventions: Device: MicroNet covered stent implantation in the increased risk arterial lesions beyond the carotid bifurcation

INTERVENTIONS:
Device: MicroNet covered stent implantation in the increased risk arterial lesions beyond the carotid bifurcation — Implantation of the MicroNet covered stent in the increased risk arterial lesions beyond the carotid bifurcation as per Vascular Team recommendation

SUMMARY:
Prospective observational study of MicroNet covered stent implantation in the elevated risk peripheral lesions (high lesion load, thrombus containing, highly calcified).

Open-label, non randomized, single arm observational study. Jagiellonian University Medical College research project.

DETAILED DESCRIPTION:
Peripheral artery stents in routine use (both balloon expandable and self-expendable) do not sufficiently prevent distal embolization. They might induce a "cheese-grater" effect - a consequence of their single layer design with uncovered space between stent struts.

Aim of the study is to evaluate short and long term safety and efficacy of MicroNet covered stent implantation in the high risk lesions beyond the carotid bifurcation. Treatment eligibility will be evaluated by a Vascular Team process (angiologist, vascular surgeon, cardiologist). Optimal pharmacotherapy will be administered according to the current guidelines.

Symptomatic and asymptomatic patients with peripheral artery disease requiring endovascular treatment for high risk stenosis (soft plaque, highly calcific plaque) per Vascular Team assessment.

A group of 30-50 consecutive patients meeting inclusion and exclusion criteria will be enrolled.

ELIGIBILITY:
General

Inclusion Criteria:

* Patients older than 18 years, eligible for peripheral artery stenting after Vascular Team evaluation, according to local standards
* Written, informed consent to participate
* Agreement to attend protocol required (standard) follow up visits and examinations

Exclusion Criteria:

* Life expectancy <1 year (e.g. active neoplastic disease).
* Chronic kidney disease with creatinine > 3.0 mg/dL.
* Myocardial infarction in 72 hours proceeding the stenting procedure (if possible, postponing the procedure)
* Pregnancy (positive pregnancy test)
* Coagulopathy.
* History of uncontrolled contrast media intolerance

Angiographic

Inclusion Criteria:

* De novo lesion in major arteries or grafts connecting arteries
* Stenosis eligible for endovascular treatment per Vascular Team evaluation (according to current standards and guidelines)
* High risk morphology stenosis (per 2 independent, experienced operators)

Exclusion Criteria:

* Chronic total occlusion not amenable to re-canalization
* Stent in the target vessel/lesion
* Anatomic variants precluding stent implantation
* Mobile (free-floating) plaque elements in aorta or arteries proximal to target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral artery stenosis evaluated by Vascular Team with endovascular treatment recommendation and high risk morphology plaque
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of procedural success | Up to 48 hours after procedure or until hospital discharge, whichever came first.
  Procedural success, defined as technical success (successful delivery and implantation of the stent) AND residual stenosis ≤ 30% of vessel lumen diameter AND clinical success (no peri-procedural complications)

SECONDARY OUTCOMES:
Number of In-hospital MACNE (Major Adverse Cardiovascular or Neurological Events) | Up to 48 hours after procedure or until hospital discharge, whichever came first.
  In-hospital MACNE (death, stroke, myocardial infarction, acute limb or target organ ischemia)
Number of MACNE at 30 days | At 30 days after procedure
  MACNE at 30 days (death, stroke, myocardial infarction, acute limb or target organ ischemia)
Number of MACNE at 6 months | At 6 months after procedure
  MACNE at 6 months (death, stroke, myocardial infarction, acute limb or target organ ischemia)
Rate of peri-procedural complications | Up to 48 hours after procedure
  Any peri-procedural complications until 48 hrs
Duplex Ultrasound Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) in the stented segment at discharge | 24 hours after procedure
  Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) on ultrasound evaluation of the stented segment (if accessible)
Duplex Ultrasound Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) in the stented segment at 6 months | At 6 months after procedure
  Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) on ultrasound evaluation of the stented segment (if accessible)
Duplex Ultrasound Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) in target vessel at 12 months | At 12 months after procedure
  Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) on ultrasound evaluation of the stented segment (if accessible)
Vessel patency in CT angiography at 6 months | At 6 months after procedure
  Vessel patency in CT angiography (if not contraindicated) at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Musialek, MD, DPhil, Principal Investigator — John Paul II Hospital, Krakow
Locations (1):
- Department of Cardiac and Vascular Diseases, The John Paul II Hospital, Krakow, Maloplska, Poland